CLINICAL TRIAL: NCT03007264
Title: Safety Assessment of Cold Gas Plasma on Intact Skin
Brief Title: Cold Plasma for Wound Treatment, Safety Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Association of Dutch Burn Centres (Other)
Collaborators: Eindhoven University of Technology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NBS 14.200-CAP1; NL52211.094.16 (Other: ABR)
Record Dates: First submitted 2016-12-23; First posted 2017-01-02 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2018-06

CONDITIONS: Intact Skin; Contaminant Given to Patient
Keywords: cold atmospheric plasma; pain; bacteria; skin parameters
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CAP treated (Experimental): volar arm will be treated with cold atmospheric plasma.
  Interventions: Device: Cold Atmospheric Plasma
- CAP on bacteria (Experimental): volar arm with bacteria will be treated with cold atmospheric plasma.
  Interventions: Device: Cold Atmospheric Plasma
- no CAP on bacteria (No Intervention): volar arm with bacteria will not be treated with cold atmospheric plasma. Sham comparator for measurements of skin parameters TEWL, temperature and bacterial load.

INTERVENTIONS:
Device: Cold Atmospheric Plasma — CAP will be applied on one volar arm of volunteers for a total of 2 minutes.
  Arms: CAP on bacteria; CAP treated

SUMMARY:
In this study the application of cold atmospheric plasma (CAP) will be tested on intact skin of volunteers. To test safety, several skin parameters will be monitored, the antimicrobial effect will be investigated as well. The investigators expect this treatment to have a good antimicrobial effect with acceptable, transient skin sensations.

DETAILED DESCRIPTION:
Control of infection and bacterial colonisation constitutes a continuing challenge in patients with burns. Prevention of microbial contamination and infection is vital for burn wound care as bacterial presence can result in excessive inflammatory reactions, delayed re-epithelialisation, impaired matrix remodelling and bacteraemia. A novel method to decrease the likelihood of infection and to help cure wounds is cold atmospheric plasma (CAP). CAP has been shown in vitro to kill a wide range of pathogenic bacteria.

This safety study aims to demonstrate the safety, efficacy and efficiency of CAP for burn wound treatment. Intact skin of volunteers will be CAP treated. Local skin reaction (blister formation, pain, itching), erythema, local skin temperature, trans epidermal water loss (TEWL) and reduction of the bacterial load wil be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to comply with the research protocol
* No language barrier

Exclusion Criteria:

* Atopic dermatitis or other skin disease
* Implanted electrical medical devices such cardiac pacemakers
* Pregnant or lactating women
* Patients with infected wounds.
* Life-threatening cardiac conductivity abnormality
* Active malignancy
* Women of childbearing age not using contraceptive measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2018-07-12 (Actual); Study Completion 2018-07-26 (Actual)

PRIMARY OUTCOMES:
pain | before to 30 minutes after treatment
  by using a visual analogue thermometer (VAT)

SECONDARY OUTCOMES:
local skin reaction | directly to 30 minutes after treatment
  blister formation, itching
local skin temperature | before to 30 minutes after treatment
  thermographic analysis
colour/pigmentation | before to 30 minutes after treatment
  erythema, redness of the skin, by using a Dermaspectrometer
trans epidermal water loss | before to 30 minutes after treatment
  barrier function of the skin by using TEWAmeter
reduction of the bacterial load | directly to 5 minutes after treatment
  quantified with scrub wash method

CONTACTS AND LOCATIONS:
Overall Officials: Esther Middelkoop, PhD, Principal Investigator — Red Cross Hospital
Locations (1):
- Association of Dutch Burn Centres, Beverwijk, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kisch T, Schleusser S, Helmke A, Mauss KL, Wenzel ET, Hasemann B, Mailaender P, Kraemer R. The repetitive use of non-thermal dielectric barrier discharge plasma boosts cutaneous microcirculatory effects. Microvasc Res. 2016 Jul;106:8-13. doi: 10.1016/j.mvr.2016.02.008. Epub 2016 Mar 2. PMID 26944583
- [Result] Brehmer F, Haenssle HA, Daeschlein G, Ahmed R, Pfeiffer S, Gorlitz A, Simon D, Schon MP, Wandke D, Emmert S. Alleviation of chronic venous leg ulcers with a hand-held dielectric barrier discharge plasma generator (PlasmaDerm((R)) VU-2010): results of a monocentric, two-armed, open, prospective, randomized and controlled trial (NCT01415622). J Eur Acad Dermatol Venereol. 2015 Jan;29(1):148-55. doi: 10.1111/jdv.12490. Epub 2014 Mar 25. PMID 24666170